CLINICAL TRIAL: NCT04630678
Title: Individualized Virtual Reality in the Upper Extremity Rehabilitation of Hemiparetic Cerebral Palsy: an Evaluator Blinded, Randomized Controlled Study
Brief Title: Individualized Virtual Reality in the Upper Extremity Rehabilitation of Hemiparetic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Mert Doğan, Master of Science, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/08-23, KA-17050
Record Dates: First submitted 2020-11-07; First posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Cerebral Palsy, Spastic
Keywords: Cerebral Palsy; Upper Extremity Rehabilitation; Virtual Reality; Technology-Assisted Therapy,; Active Video Game
MeSH Terms: conditions — Cerebral Palsy | interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Intervention Model Description: The children were randomized into two groups.The first group was received virtual reality therapy. The second group was received activity training. Both treatments were given three times a week for eight weeks.
Who Masked: Outcomes Assessor
Masking Description: The children in both groups were evaluated by the same physiotherapist who was blinded. The treatment was given by a different physiotherapist who has been working in the field of pediatric physiotherapy for ten years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): The first group was received conventional physiotherapy and virtual reality therapy for 60 minutes.
  The conventional physiotherapy interventions, including joint and muscle mobilization, strengthening, and stretching exercises by neurodevelopmental treatment principles and special for the needs of the child, was applied to both groups. The virtual reality group received that simulate daily life and contain individual scenarios by using the USE-IT system for thirty minutes. USE-IT (Most Rehabilitation, Ankara, Turkey) is a 2D non-immersive virtual reality system that plays games on a 50-inches touchscreen. The children played "the matching, plumber, plumber, math, and car wash games" in accordance with their reaching map results. The treatment were given three times a week for eight weeks.
  Interventions: Other: Virtual Reality Therapy; Other: Conventional Physiotherapy
- Activity Training (Control) Group (Active Comparator): The second group was received conventional physiotherapy and, activity training which the same movement patterns with virtual reality games for 60 minutes. The children in the activity training group received unilateral, bilateral, and bimanual activity training that supported manual skills for thirty minutes. Similar activity patterns were presented to the virtual reality group and activity training (control) group. The treatment were given three times a week for eight weeks.
  Interventions: Other: Conventional Physiotherapy; Other: Activity Training

INTERVENTIONS:
Other: Virtual Reality Therapy — Virtual reality games were applied to participants for 30 minutes.
  Arms: Virtual Reality Group
Other: Conventional Physiotherapy — Joint and muscle mobilization, strengthening, and stretching exercises by neurodevelopmental treatment principles were applied to participants for 30 minutes.
Other: Activity Training — Unilateral, bilateral, and bimanual activity training that supported manual skills for 30 minutes.
  Arms: Activity Training (Control) Group

SUMMARY:
This study aimed to investigate the effect of individualized virtual reality therapy on upper extremity functions of children with hemiparetic cerebral palsy.

Forty children (26 boys, 14 girls) with spastic hemiparetic cerebral palsy were included in this study. The primary outcome measure of this study was the Quality of Upper Extremity Skill Test, secondary outcome measures were the Modified Ashworth Scale and the "Reaching Map Test". The children were randomized into two groups. The first group was received conventional physiotherapy and virtual reality therapy for 60 minutes.The second group was received conventional physiotherapy and, activity training which the same movement patterns with virtual reality games for 60 minutes. Both treatments were given three times a week for eight weeks.

DETAILED DESCRIPTION:
Participants Forty children (20 boys, 20 girls) were included in the study, and their demographic information was recorded. The participants were divided, using "randomizer.org" with a simple randomization method, into two different groups: the Virtual Reality or Activity Training (control) groups.

Study Design All children were assessed at baseline and after eight weeks of treatment. The children in both groups were evaluated by the same physiotherapist who was blinded. The treatment was given by a different physiotherapist who has been working in the field of pediatric physiotherapy for ten years Interventions The participants were randomized into two groups. The first group was received conventional physiotherapy and virtual reality therapy for 60 minutes. The second group was received conventional physiotherapy and, activity training which the same movement patterns with virtual reality games for 60 minutes. Both treatments were given three times a week for eight weeks.

The conventional physiotherapy interventions, including joint and muscle mobilization, strengthening, and stretching exercises by neurodevelopmental treatment principles and special for the needs of the child, was applied to both groups. The virtual reality therapy group received that simulate daily life and contain individual scenarios by using the USE-IT system for thirty minutes. USE-IT (Most Rehabilitation, Ankara, Turkey) is a 2D non-immersive virtual reality system that plays games on a 50-inches touchscreen. The children played "the matching, plumber, plumber, math, and car wash games" in accordance with their reaching map results. As the system detects not only hand but also object touch the real-life materials (cloths and hoses etc.) were used to stimulate grip and sense during games. The children in the activity training group received unilateral, bilateral, and bimanual activity training that supported manual skills for thirty minutes. Similar activity patterns were presented to the virtual reality group and activity training group.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as spastic hemiparetic cerebral palsy by a physician,
* must be level I, II, and III according to the Gross Motor Function Classification System (GMFCS)
* must be level I, II, and III according to the Manuel Ability Classification System (MACS)

Exclusion Criteria:

* have cardiac or orthopedic contraindications for sitting, standing, and walking
* have orthopedic surgery to upper extremity and trunk in the last 6 months
* have used of spasticity-reducing medication or botulinum toxin injections to upper extremity or trunk in the last 6 months
* being severely mentally affected
* have any neurological conditions accompanying cerebral palsy (seizures, visual deficits, etc.)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline "The Quality of Upper Extremity Skills Test Scores" at 8 weeks. | At baseline and after 8 weeks treatment.
  The Quality of Upper Extremity Skills Test was used to assess the function and quality of upper limb movements. This test has a total of 7 subdivisions, and the scoring of each section is calculated using a standardized formula. Each chapter is scored between 0-100 within itself. The first four section scores are used to calculate the total score. A high score indicates better the quality of the movement. The participant evaluated by a physiotherapist at baseline and after 8 weeks treatment.

SECONDARY OUTCOMES:
Change from Baseline "The Modified Ashworth Scale Scores" at 8 weeks. | At baseline and after 8 weeks treatment.
  The Modified Ashworth Scale was used to assess the severity of spasticity of shoulder internal rotators, elbow, wrist, and finger flexors and elbow pronators, thumb abductors. The score is between 0-5 for each muscle. As the score increases, the severity of spasticity increases.
Change from Baseline "The Reaching Map Test Scores" at 8 weeks. | At baseline and after 8 weeks treatment.
  Forty balloons, randomized, appears on the screen, and the system asked the child to exploded the balloons. The child was positioned in front of the screen, and hip-knee angles were positioned 90° flexion. Through the special algorithm in the system, the "individual" access area was determined, and the scenario of the games was automatically adjusted accordingly. The areas that the child can reach on the screen were divided into five difficulty levels. Five levels from easy to very difficult describe as yellow, green, blue, navy blue and red areas were automatically calculated by the USE-IT system.

CONTACTS AND LOCATIONS:
Overall Officials: Mert Doğan, mSc, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No